CLINICAL TRIAL: NCT07072715
Title: The Effectiveness of Plyometric Training and Post-Activation Performance Enhancement Intervention on Agility, Explosive Power, and Speed in Football Players: A Randomized Controlled Trial
Brief Title: Plyometrics vs PAPE Training in Football: Effects on Agility, Explosive Power and Speed
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Yassmin Ibrahim Talaat Badr, Master's Student Researcher, Istinye University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-87
Record Dates: First submitted 2025-07-08; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Athletic Performance; Football Players; Sports Performance; Sports Physical Therapy
MeSH Terms: interventions — Plyometric Exercise

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PAPE Training Group (Experimental): Participants in this group received post-activation performance enhancement (PAPE) training using high-resistance banded squats (~85% 1RM) 3 times per week for 8 weeks, immediately after warm-up and before continuing their regular football training. 10% of load was added every week to their training load. 3 reps and 3 sets were done per session with 5 minutes of active rest interval between sets.
  Interventions: Behavioral: PAPE Training
- Plyometric Training Group (Experimental): Participants in this group performed additional plyometric training 3 times per week for 8 weeks, immediately after warm-up and before continuing their regular football training. Training included depth jumps using a plyometric box with gradual increase in height of the box from 30-60 cm. 12 reps and 7 sets were performed with 30 seconds- 1 minute of rest interval between sets
  Interventions: Behavioral: Plyometric Training
- Control Group (No Intervention): Participants in this group continued with their regular football training routine without receiving any additional intervention.

INTERVENTIONS:
Behavioral: PAPE Training — A neuromuscular activation protocol involving heavy banded squats (~85% 1RM) to induce post-activation performance enhancement. Applied three times weekly over 8 weeks following the warm-up. Participants then continued with regular football training.
  Other Names: Post Activation Performance Enhancement Training
  Arms: PAPE Training Group
Behavioral: Plyometric Training — A program of depth jumps designed to enhance explosive power, speed, and agility. Applied 3 times weekly over 8 weeks following the warm-up. Participants then continued with their regular football training.
  Arms: Plyometric Training Group

SUMMARY:
The goal of this clinical trial is to compare the effects of 8 week plyometric training and post-activation performance enhancement (PAPE) training on explosive power, agility, acceleration and sprint speed, muscle strength and flexibility in healthy male semi-professional football players aged 18-35.

The main questions it aims to answer are:

Does PAPE training have effects on performance metrics of football players when planned and applied long-term (8 weeks)?

Does long term PAPE training improve agility, acceleration and speed, flexibility, vertical jump height, and muscle strength more effectively than Plyometric training?

Is there a significant difference in performance gains between PAPE and plyometric training compared to a control group receiving only routine football training?

Researchers will compare a plyometric training group, a PAPE training group, and a control group to determine which method most effectively enhances football-specific performance outcomes.

Participants will:

* Be randomly assigned to one of three groups (Plyometric, PAPE, or Control)
* Continue their routine football training as usual
* Receive additional training sessions applied immediately after warm-up and before continuing regular team training alongside the Control group (for PAPE and Plyometric group)
* Undergo an 8-week training program (3 times per week for Plyometric and PAPE groups)

Assessments will be conducted at baseline, week 4, and week 8, including:

* Vertical Jump Test (explosive power)
* 30-Meter Sprint Test, including 10-meter acceleration recording
* Illinois Agility Test
* Isometric strength measurements of quadriceps, hamstrings, and gastrocnemius using a handheld dynamometer
* Sit and Reach Test and Modified Thomas Test (flexibility)

In addition, all participants will complete a sociodemographic and lifestyle assessment form capturing:

Age, height, weight, BMI Football experience and playing position Education level, employment status Sleep duration, training frequency, and training intensity Smoking and alcohol use status.

ELIGIBILITY:
Inclusion Criteria:

* Male athletes aged between 18 and 35 years
* Permission obtained from the team physician to participate in the study
* Active participation in a Semi-Professional football team for at least the past 6 months
* Participating in football training at least 3 times per week
* Willing and able to participate in 8-week training and testing protocol voluntarily

Exclusion Criteria:

* Current or recent surgery affecting the lower limbs
* Current or recent injury affecting the lower limbs
* History of neurological, cardiovascular, orthopedic or systemic disease
* Inconsistent football training (<3x per week)
* Failure to attend testing or training sessions

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Illinois Agility Test | Baseline, Week 4, Week 8
  Time to complete the Illinois Agility Test will be measured under standardized conditions with a stopwatch. Participants sprint and weave through cones in a pre-set course. The total time to complete the course is recorded; best of two attempts is used.
Vertical Jump Height (Countermovement Jump) | From Baseline to Week 4 through Week 8
  Vertical jump height will be assessed using the "MyJump 2" app specifically the Counter Movement Jump with Free Arms (CMJ). A video of the participant will be taken and using frame selection of take-off and landing, their jump height will be automatically calculated by the app. Three attempts will be averaged.
30-Meter Sprint Time (including 10-meter split) | Baseline, Week 4, Week 8
  Sprint time over 30 meters will be recorded using stopwatch with a 10-meter acceleration split included.
Vertical Jump Test (Sargent Jump) | Baseline, Week 4, Week 8
  Vertical jump height will be measured using the Sargent Jump Test, a standardized field-based assessment of lower-body explosive power. Participants will stand adjacent to a wall, reach up to mark their standing reach height, then perform a maximal vertical jump and touch the wall at the peak of the jump. The difference between the standing reach and jump reach (in centimeters) will be recorded as the jump height. Each participant will perform three trials, and the average will be used for analysis.

SECONDARY OUTCOMES:
Isometric Muscle Strength (Quads, Hamstrings, Gastrocnemius) | Baseline, Week 4, Week 8
  Maximal voluntary isometric contraction will be measured using a handheld dynamometer across three muscle groups for both left and right sides of the lower extremity. Mean of three trials per muscle group will be used.
Sit and Reach Test | Baseline, Week 4, Week 8.
  Measures hamstring and lower back flexibility using a sit-and-reach box. Participants perform three attempts; the best distance reached (in cm) is recorded.
Modified Thomas Test | Baseline, Week 4, Week 8.
  Hip flexor and quadriceps flexibility are assessed using the Modified Thomas Test with goniometric measurement. Angles are recorded in degrees; each leg is tested once.

OTHER OUTCOMES:
Sociodemographic and Lifestyle Profile | Baseline only (Week 0)
  Participants will complete a structured questionnaire at baseline to collect data on age, height, weight, BMI, football experience (in years), playing position, education level, employment status, sleep duration, training frequency and intensity, and smoking/alcohol use.
  This information may be used for exploratory subgroup or correlational analyses to examine its potential influence on performance outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Habibe S. Inal, Prof. Dr, Principal Investigator — Galata University
Locations (1):
- Fatih Karagümrük A.Ş., Istanbul, Turkey (Türkiye)